CLINICAL TRIAL: NCT03228628
Title: Impact of 50% Nitrous Oxide Inhalation on Pain and Anxiety Induced by Lumbar Puncture: a Multicenter Double-blind Randomized Controlled Trial
Brief Title: Nitrous Oxide for Lumbar Puncture
Acronym: NO for LP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Bordeaux (Other); Hospices Civils de Lyon (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-342; 2017-002750-37 (Other: 2017-002750-37)
Record Dates: First submitted 2017-07-19; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Pain; Anxiety
Keywords: Spinal puncture; Pain; Anxiety; Nitrous oxyde
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to receive experimental treatment (50% N2O - 50% O2) or placebo (Medical Air: 22% O2 - 78% N2)
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinding. Gaz bottles are in undistinguishable boxes. Neither the patients nor the person doing the LP and the evaluation of pain and anxiety will know the treatment used
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrous oxide (Experimental): will inhale experimental treatment (50% N2O - 50% O2)
  Interventions: Drug: Fixed 50:50 mixture of nitrous oxide and oxygen
- Placebo (Placebo Comparator): will inhale medical air (22% O2 - 78% N2)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fixed 50:50 mixture of nitrous oxide and oxygen — Gaz inhalation will start 5 minutes before the puncture and will be continued until the end of the procedure.
  Arms: Nitrous oxide
Other: Placebo — inhale medical air (22% O2 - 78% N2)
  Arms: Placebo

SUMMARY:
Lumbar puncture (LP) is a frequent exam that can cause pain and anxiety. In a pilot single-center study, it has been shown that nitrous oxide use during the procedure was able to reduce both pain and anxiety (Moisset et al., Eur J Neurol 2017). The goal of this multi-center trial is to confirm these results in a larger and more heterogeneous group of patients having a LP.

DETAILED DESCRIPTION:
Nitrous oxide (N2O) has analgesic and anxiolytic properties that are known for more than a century. Nonetheless, it's use during lumbar puncture in adults has only been investigated in a single-centre study.

Thus, this study is designed to evaluate the analgesic effect of N2O on the pain induced during lumbar puncture.

Patients with scheduled lumbar puncture realized for diagnosis purposes will be randomized in 2 groups. One group will inhale N2O for the 5 minutes before the puncture and during the rest of the procedure. The second group will inhale compressed air during the same period of time. Neither the investigator realizing the lumbar puncture, nor the patient will know which type of gaz they are inhaling (double-blinding).

The maximal pain level that occurred during the procedure will be evaluated on a Numerical Rating Scale (NRS). NRS will also be used to evaluate the maximal anxiety induced by the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients coming in the neurology department for a lumbar puncture
* at least 18
* no previous use of nitrous oxide

Exclusion Criteria:

* contra-indication to nitrous oxide use
* Body Mass Index>35
* Mini Mental State Examination <24/30
* Temperature >38°C
* Confusion
* Patient unable to communicate verbaly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-06-06 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with significant pain | 2-3 minutes after the end of gaz inhalation
  maximal pain perceived during the lumbar puncture evaluated using a simple numeric 0-10 pain scale

SECONDARY OUTCOMES:
Proportion of patients with significant anxiety | 2-3 minutes after the end of gaz inhalation
  maximal anxiety perceived during the lumbar puncture evaluated using a simple numeric 0-10 scale
Analgesic efficacy measured with pain as a continuous variable | 2-3 minutes after the end of gaz inhalation.
  maximal pain perceived during the lumbar puncture evaluated using a simple numeric 0-10 pain scale
Anxiolytic efficacy measured with anxiety as a continuous variable | 2-3 minutes after the end of gaz inhalation
  maximal anxiety perceived during the lumbar puncture evaluated using a simple numeric 0-10 scale
Pain during the procedure evaluated one hour after the end of the lumbar puncture | 1 hour after the end of gaz inhalation
  maximal pain and anxiety perceived during the lumbar puncture evaluated using a simple numeric 0-10 scale
Anxiety during the procedure evaluated one hour after the end of the lumbar puncture | 1 hour after the end of gaz inhalation
  maximal pain and anxiety perceived during the lumbar puncture evaluated using a simple numeric 0-10 scale
Side effects | from the beginning of gaz inhalation to 24 hours later
  every side effects reported by the patients during the procedure up to 24 hours after the lumbar puncture, including post-puncture puncture headache
Impact of age on side effects | during the procedure and the 24 hours after
  incidence and type of side effects according to patient age
Induced cost | at day 1
  supplementary cost induced by the use of nitrous oxide inhalation for a total of 81 patients throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MOISSET, MD-PhD, Principal Investigator — CHU Clermont-Ferrand, Inserm, Neuro-Dol
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France